CLINICAL TRIAL: NCT03044756
Title: Impact of Omitting GnR-antagonist on Ovulation Trigger Day in the Fresh Autologous IVF/ICSI Cycles
Brief Title: Omitting GnRH-antagonist Dose on the Day of Ovulation Trigger
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Lecturer of OBGYN, Women Health Hospital, Assiut Univerisity, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Omit
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Pituitary Downregulation
Keywords: GnRH antagonist; Pituitary downregulation; IVF; ICSI

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- -ve arm (Experimental): The women who do not receive the GnRH antagonist dose on the day of triggering of ovulation (omitted GnRH antagonist arm)
  Interventions: Drug: Omit Citrotide 0.25 dose on the day of triggering of ovulation
- +ve arm (No Intervention): The women who receive the routine dose of GnRH antagonist on the day of triggering of ovulation (the usual protocol)

INTERVENTIONS:
Drug: Omit Citrotide 0.25 dose on the day of triggering of ovulation — Omit Citrotide 0.25 dose on the day of triggering of ovulation
  Arms: -ve arm

SUMMARY:
Omitting the GnRH antagonist on the day of the trigger can be cost effective and more convenient to the women. We will study the impact of omitting the antagonist dose in a prospective randomized trial

ELIGIBILITY:
Inclusion Criteria:

* All antagonist cycle ivf who agree to participate

Exclusion Criteria:

* expected poor responders.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved oocytes | One Month
  total number and maturation of the retrieved oocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Osama Abdalmageed, Asyut, Non-US/Non-Canadian, Egypt

IPD SHARING:
Plan to Share IPD: No
The regulations in Assiut University do not allow protected patient data sharing

REFERENCES:
- [Background] Chang HJ, Lee JR, Jee BC, Suh CS, Lee WD, Kim SH. Cessation of gonadotropin-releasing hormone antagonist on triggering day in flexible multiple-dose protocol: A randomized controlled study. Clin Exp Reprod Med. 2013 Jun;40(2):83-9. doi: 10.5653/cerm.2013.40.2.83. Epub 2013 Jun 30. PMID 23875164